CLINICAL TRIAL: NCT05484180
Title: The Effect of Guided Imagery Based on the Health Promotion Model on the Quality of Life in Breast Cancer Patients: An Integrative Study
Brief Title: The Effect of Guided Imagery Based on the Health Promotion Model on the Quality of Life in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülnaz Ata, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Glnz87?
Record Dates: First submitted 2022-07-24; First posted 2022-08-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer Female
Keywords: Guided Imagery; Breast Cancer; Nursing; Quality of Life; Healthy Lifestyle Behaviors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization was done with 68 people. Simple randomization method was used in order to assign 68 people included in the study to the experimental and control groups in an unbiased manner. For randomization, a sample pool of people included in the study was created. Randomization was done in computer environment using https://www.random.org/ website. The women in the experimental and control groups were determined according to the order obtained. In this way, 34 individuals were included in the experimental group and 34 individuals in the control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the data collection process, double-blindness was provided by not specifying which group the interviewer was collecting data from and which group participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): As a nursing initiative to the experimental group in the research; Training and consultancy supported guided imagery application based on the health promotion model was applied.
  Interventions: Other: training and counseling supported guided imagery application
- control group (No Intervention): No attempt will be made on individuals in the control group during the research process. After the research process is over; After the training booklet, Mp3 player loaded with directed imagery recording and exercise materials are delivered, guided imagery application based on the Health Promotion Model will be supported by training and counseling.

INTERVENTIONS:
Other: training and counseling supported guided imagery application — After the preparation process, as a nursing attempt to the individuals in the experimental group; Training and consultancy supported guided imagery based on the health promotion model will be implemented. This initiative; It will take a total of 12 weeks, including 6 weeks of training program and 6 weeks of counseling program and guided imagery.
  Arms: experimental group

SUMMARY:
This research is a randomized controlled double-blind experimental study aiming to evaluate the effect of guided imagery based on the health promotion model in breast cancer patients on healthy lifestyle behaviors and quality of life. Research; It will be carried out between January-September 2022 with patients diagnosed with breast cancer who have completed the treatment process and registered in the Medical Oncology Polyclinic of Ataturk University Health Research and Application Center. The sample of the study will consist of 70 people, 34 of which are in the experimental group and 34 in the control group. After obtaining verbal and written consents from all sampled individuals, respectively; Introductory Information Form, Healthy Lifestyle Behaviors Scale II, SF-36 Quality of Life Scale and Body Mass Index Assessment will be applied as pre-test. Then, as a nursing attempt to the individuals in the experimental group; Training and consultancy supported guided imagery based on the health promotion model will be implemented. This initiative; It will take a total of 12 weeks, including 6 weeks of training program and 6 weeks of counseling program and guided imagery. After the application is completed, post-test measurements of the patients in the experimental and control groups will be made. For final test measurements; Healthy Lifestyle Behaviors Scale II, SF-36 Quality of Life Scale and Body Mass Index Assessment will be performed; Feedback will be received from the patients in the experimental group regarding the research process. No attempt will be made to the individuals in the control group during the research process, and after the research process is over, the same intervention applied to the experimental group will be applied to the control group. Then, the feedback of the individuals in the control group regarding the research process will be received. The data obtained in the research will be evaluated in the SPSS 22.00 package program. Ethical principles will be followed at all stages of the research, for which ethics committee approval has been obtained, and the Helsinki Declaration of Human Rights will be adhered to. It is planned to present the results of the research at an international congress and to be published in a journal within the scope of SCI/SSCI, to be brought to the scientific literature and announced.

Keywords: Breast Cancer, Guided Imagery, Health Behaviors, Health Promotion Model, Nursing, Quality of Life

DETAILED DESCRIPTION:
İntroduction Breast cancer; It is an important public health problem because it is the most common cancer type globally and is closely associated with mortality. Breast cancer, which is a chronic disease and continues throughout life; It negatively affects many aspects of life with its individual, familial and social dimensions. Due to both the disease and a long and difficult treatment process, many individual and social changes are experienced in the process after the active treatment of breast cancer is completed, physical discomforts such as fatigue and pain continue, and many problems such as fear of recurrence of the disease and changes in body image occur in life quality and well-being are significantly affected. In addition, in this process, patients; They may experience many problems such as permanent side effects of the treatment, stress and depression, and they need to be informed about lifestyle changes.

Despite that; When the literature is examined, while the problems of cancer patients during the treatment process are considered more important, they are not given enough attention after the treatment process and there are limited number of studies on the problems experienced in this period. At this point, studies based on the Health Promotion Model, which include the processes of acquiring health promoting behaviors in detail and which is one of the most widely used models in nursing research, are of great importance. According to the literature, healthy lifestyle behaviors prevent late problems, chronic disease risks, recurrences, secondary cancers and reduce mortality in cancer patients; on the other hand, it is stated that it increases individual coping and quality of life, supports the individual holistically, and reduces health expenditures. One of the most used integrative/holistic applications in cancer patients today is guided imagery. In addition to contributing to the development of targeted behavior, guided imagery; by making the patient's mind get away from disturbing emotions and negative thoughts in daily life and feel relaxed, happy and peaceful; positively affects well-being, self-efficacy and quality of life. As it is known, the quality of life is one of the United Nations Sustainable Development Goals and is considered internationally important. When the literature is examined, guided imagery has been applied in cancer patients, especially for the management of symptoms such as pain, fatigue, nausea-vomiting, insomnia, stress and anxiety, in individuals whose treatment process is ongoing. No study was found that evaluated the simultaneous effects of the health promotion model and guided imagery. A guided imagery method that positively supports individuals' well-being and quality of life by providing mind-body harmony.

Keywords: Breast Cancer, Health Promotion Model, Guided Imagery, Nursing, Quality of Life, Healthy Lifestyle Behaviors

Research Hypotheses H1a: After the training and counseling supported guided imagery application based on the health promotion model in the experimental group, the healthy lifestyle behaviors mean scores of the participants were higher than before the application (within group) and control group (between groups).

H1b: After the training and counseling supported guided imagery application based on the health promotion model in the experimental group, the health-related quality of life score averages of the participants were higher than before the application (within group) and control group (between groups).

This research is a randomized controlled experimental study aiming to evaluate the effect of education and counseling supported guided imagery application based on the health promotion model in breast cancer patients on healthy lifestyle behaviors and quality of life.

Research; It will be carried out between 01 February 2022 and 01 February 2023 with individuals diagnosed with breast cancer who have completed the treatment process and reside in Erzurum city center, registered in the Medical Oncology Polyclinic of Atatürk University Health Research and Application Center.

Population and Sample of the Research The universe of the research; consists of individuals with breast cancer who have completed the treatment process and reside in Erzurum city center and are registered to the relevant oncology outpatient clinic (N=291). The sample number is; Similar studies in the G*Power 3.1 program were calculated as, taking into account 50% effect size, 95% reliability and 95% theoretical power. However, it was determined that 70 people would be included in the study by adding 16 people (30% more than the sample number) to the determined sample, in case the participants could withdraw from the study at any stage of the research. The systematic sampling method was used to determine the 70 people to be sampled. The women selected from the list by systematic sampling method were called by phone, informed about the research and invited to the research. Those who agreed to participate in the study were included in the sample after obtaining their verbal consent from those who met the inclusion criteria. If the sample size could not be reached due to reasons such as the criteria were not met or the research invitation was not accepted, the systematic sampling method was repeated within the same list until the targeted sample size was reached.

In the pre-test phase of the research, two people left the study voluntarily. For this reason, randomization was made with 68 people. A simple randomization method was used in order to assign people included in the study to the experimental and control groups in an unbiased manner. Randomization was done in computer environment using https://www.random.org/ website. The women in the experimental and control groups were determined according to the order obtained. In this way, 34 individuals were included in the experimental group and 34 individuals in the control group. After randomization, the homogeneity of the groups according to the control variables was evaluated and the groups were found to be homogeneous.

Variables of the Study Dependent variables: Healthy lifestyle behaviors, quality of life. Independent variables: Guided imagery practice, training and counseling program.

Control variables: Age, education level, childbearing status, time of diagnosis of disease, clinical stage diagnosed, treatment completed.

Data Collection Tools In the collection of research data; Introductory Information Form, Healthy Lifestyle Behaviors Scale II and SF-36 Quality of Life Scale will be used. In addition, the Body Mass Index (BMI) of all participants will be evaluated. In the research, the "Feedback Form on the Research Process" will be applied to all participants.

Data Collection Pre-test and post-test data of the research; After obtaining written consent from the individuals included in the study, it was collected face-to-face by an interviewer who was pursuing his graduate education in public health nursing and was trained in the research process and data collection process. In the data collection process, double-blindness was ensured by not telling the interviewer from which group the data was collected and which group they were in.

Pre-Test Data Collection Experiment and control groups in the pre-test; Introductory Information Form, Healthy Lifestyle Behaviors Scale II and SF-36 Quality of Life Scale were applied and BMI Evaluation was made. Data collection took an average of 45 minutes for each individual, and the data were collected face-to-face by the interviewer during a home visit. Pre-test data were collected between 04 April 2022 and 23 May 2022.

Collection of Post-Test Data After the training and counseling supported guided imagery application based on the health promotion model was completed, in the collection of post-test data, individuals in the experimental and control groups; Healthy Lifestyle Behaviors Scale II and SF-36 Quality of Life Scale will be applied and BMI Assessment has been made. In addition, the participants in the experimental group regarding the research process were evaluated with the "Research Process Feedback Form". Data collection took an average of 45 minutes for each individual. The data were collected face-to-face by the interviewer during a home visit. It is planned to collect post-test data between 22 August and 15 September 2022.

Pilot Application In the research; A pilot study was conducted on five patients who had the same characteristics as the sample group but who would not be included in the main study.

Nursing Interventions As a nursing initiative to the experimental group in the research; Training and consultancy supported guided imagery application based on the health promotion model was applied.

Before starting any intervention, pre-test measurements of 68 individuals in the experimental and control groups were made. After the pre-test data were collected, the individuals in the experimental group were visited by the researcher at their homes; One training booklet, Mp3 player with guided imagery recording, pilates band and 0.5 kg dumbbells were delivered. Two WhatsApp groups were created separately for the experimental and control groups, and the participants were added to these groups. In addition, an e-mail address was provided to the participants. To provide an additional option for the participants regarding the accessibility of the initiative materials and to increase their permanence; The training booklet and the guided imagery recording were also sent to the individuals in the experimental group via WhatsApp to their phones and e-mails. Then, a "Google Meet" record was created for each participant. Information was given on how to use the application and how to enter the link sent via WhatsApp and e-mail. Internet support will be provided by the researcher to individuals who have internet connection problems during the research process, and this situation will be taken into account in arranging the session hours. After the preparation process, as a nursing attempt to the individuals in the experimental group; Training and consultancy supported guided imagery based on the health promotion model will be implemented. This initiative; It will take a total of 12 weeks, including 6 weeks of training program and 6 weeks of counseling program and guided imagery. After the application is completed, the post-test measurements of the individuals in the experimental and control groups will be made. No attempt will be made to the individuals in the control group during the research process. After the research process is completed, a training booklet, Mp3 player loaded with guided imagery recording, pilates tape and 0.5 kg dumbbells will be delivered to the individuals in the control group; The training booklet and the guided imagery recording will also be sent to WhatsApp and e-mails. Then the same intervention applied to the experimental group will be applied.

Educational program: The content of the training program was prepared by scanning the national and international literature and taking the opinions of four experts. Educational program; The health promotion model is based on the relationship between healthy lifestyle behaviors (nutrition, physical activity and exercise, stress management, health responsibility, interpersonal support and self-actualization) and quality of life. In addition, in the sixth week of the training program, training and information will be given about guided imagery. The training program was held with the participants at a predetermined time through the online platform "Google Meet". Since there were 34 individuals in the experimental group, the training program was carried out as group trainings in order to ensure an effective study. In this context, 34 individuals in the experimental group; Three groups of 12, 12 and 10 people attended the training sessions. The training program for each group was performed once a week and averaged 50-60 minutes each. It will consist of six sessions in total. Therefore, the training program of the experimental group will be completed in six weeks and 18 sessions in total. Oral presentation, brainstorming, question-answer, visual and subject-oriented video demonstrations, discussion and demonstration methods, powerpoint presentations and training booklets will be used in the trainings.

Counseling Program: Counseling program in research; The health promotion model will be based on the sub-components of individual characteristics and experiences, behavioral-specific cognitive factors and the emergence of behavior. Counseling program to be carried out simultaneously with the guided imagery practice; It will be held in the form of a "Google Meet" meeting for 6 weeks, in 15-day periods. The counseling program will be carried out individually, and within this scope, three "Google Meet" meetings will be held with each participant in total. These interviews last approximately 30-45 minutes. it will last. With the counseling program, reminders will be made about performing and maintaining healthy lifestyle behaviors and guided imagery to increase the quality of life of breast cancer patients, their questions will be answered, counseling will be given and follow-up will be made in line with their needs and based on the sub-components of the health promotion model.

Guided Imagery Application: In the research, guided imagery scenario content including positive directives for healthy lifestyle behaviors and quality of life was created with the support of the literature. The script content was written by Dr., who is an expert in clinical psychology and also took part in the research process as a second consultant. Instructor Prepared under the supervision of member Derya Gürcan Yıldırım. For the guided imagery scenario content prepared, expert opinions were received from 10 people from the fields of Psychiatric Nursing, Mental Health and Diseases and Clinical Psychology. Scenario content after expert opinions; It was voiced by the researcher with a musical accompaniment of relaxing, relaxing, soft and slow tempo mixed nature sounds and recorded with a voice recorder. Then the created recording was transferred to Mp3 players by the researcher. Mp3 players with guided imagery recordings were delivered to the individuals in the experimental group by the researcher after the pre-test data were collected and they were informed about their use.

Before starting the guided imagery application, the individuals in the experimental group will be told how to apply the guided imagery in the sixth week of the training program and explanations will be given before the application. In the first three days, the guided imagery application will be divided into four groups of 7 people and one of 6 people in the experimental group, divided into five groups in total by the researcher and over "Google Meet". Afterwards, the participants will be given a guided imagery application in their own homes, once a day for 6 weeks, for a period of time they have determined, accompanied by an Mp3 player loaded with the guided imagery recording delivered at the beginning of the research. At the same time, participants will be asked to record the guided imagery practice daily in the checklist on the back of the training booklet delivered at the beginning of the study. Follow-up of the participants will be made with "Google Meet" meetings in 15-day periods within the scope of the consultancy program that will be carried out simultaneously with the guided imagery application.

Evaluation of Data SPSS 22.00 package program will be used in the coding and evaluation of the data. In addition to the mean, standard deviation, numbers and percentages in the evaluation of the data, it is thought that analyzes such as t-test for independent groups, t-test for dependent groups, analysis of variance, correlation and regression analysis will be used in statistical comparisons according to the characteristics of the data. Normality distributions of the data will be evaluated with Kurtosis and Skewness coefficients, non-parametric tests will be used for data that are not normally distributed. The internal validity of the scales will be determined by the Cronbach α coefficient, and whether the descriptive features of the experimental and control groups are homogeneous will be analyzed by the chi-square test. A low p value of 0.05 will be accepted as the level of significance.

Limitations and Generalizability of the Study The limitation of the study is that the results of the study can be generalized to this group.

Ethical Principles of Research Before starting the research, approval from the Ethics Committee of Erzurum Atatürk University Faculty of Medicine and written permission from the institution where the research would be conducted were obtained. To the individuals included in the research; After the necessary explanations are made about the purpose of the research and the method of application, their verbal consent will be obtained. During the collection of research data, individuals will be informed about the research, and written consent will be obtained by following the "Informed Consent" principle, stating that they are free to participate in the research, "Respect for Autonomy", and "Confidentiality and Protection of Confidentiality" by stating that their information will be kept confidential. Those who are willing to participate in the research will be included in the research. Since individual rights must be protected in the research, the Helsinki Declaration of Human Rights will be adhered to during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed in stage I, II or III of breast cancer
* Without organ metastasis
* Those who have not been diagnosed with any other cancer other than breast cancer
* Literate
* Able to communicate verbally
* Capable of using a smartphone
* Internet connection and online access
* Those who have not practiced directed imagery before
* Declaring that they can apply the directed imagery technique
* Individuals aged 18 and over will be included in the study. Inclusion criteria will be based on the statements of individuals and patient files.

Exclusion Criteria:

* IV of breast cancer. diagnosed at stage
* Organ metastases
* Those who have been diagnosed with a cancer other than breast cancer
* illiterate
* Cannot communicate verbally
* Unable to use a smartphone
* No internet connection or online access
* Those who have practiced directed imagery before
* Individuals who declare that they cannot apply the directed imagery technique will be excluded from the sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
The sociodemographic characteristics of the participants and their homogeneous distribution according to the experimental and control groups | baseline
  The sociodemographic characteristics of the participants and their homogeneous distribution according to the experimental and control groups will be evaluated with the introductory information form. Introductory Information Form: Developed by researchers in line with the literature and prepared by taking the opinions of four experts; It includes 10 questions such as age, education level, family type, marital status, number of children, monthly income, occupation, time of diagnosis of the disease, clinical stage of diagnosis and completed treatments.
The healthy lifestyle behaviors | 12 weeks
  The healthy lifestyle behaviors of the participants will be evaluated with the Healthy Lifestyle Behaviors Scale II. The scale consists of 52 items and six sub-dimensions. The sub-dimensions of HLBD are as follows: Spiritual development, health responsibility, physical activity, nutrition, interpersonal relationships and stress management. All questions related to HLPV are weighted on a four-point Likert-type scale as never (1), sometimes (2), often (3), regularly (4). The lowest score for the whole scale is 52, and the highest score is 208.
Participants' quality of life level | 12 weeks
  The quality of life of the participants will be evaluated with the SF-36 Quality of Life Scale. The quality of life scale; It contains 36 statements that evaluate 2 main dimensions and 8 sub-dimensions. The scale has likert type scoring. 35 out of 36 statements in the scale are evaluated considering the last 4 weeks. "How do you find your current health when compared to a year ago?" which includes the perception of change in health in the last 12 months in the scale. statement is not taken into account in the evaluation. The scale does not have a single total score, and the score for each dimension is calculated separately. The scores of each sub-dimension and the two main dimensions range from 0 to 100. The positive scoring SF-36, the higher the score of each dimension; Health-related quality of life was scored as increased.
Body Mass Index (BMI) Evaluation | 12 weeks
  BMI; In the research, it will be evaluated by the interviewer twice, in the pre-test and post-test. BMI will be calculated by measuring height and weight with scales and tape measure at the participants' homes. Height and weight measurements will be made for the pre-test and post-test at the same time of the day, wearing the same clothes and taking into account the same hunger / satiety conditions. After the height and weight measurements of the participants are made, the BMI calculation will be made on the official website of the Ministry of Health. BMI; If it is less than 18.50, it will be considered as underweight, between 18.50-24.99 as normal/healthy weight, between 25-29.99 as overweight/overweight, and above 30 as overweight/obese.

SECONDARY OUTCOMES:
Feedback Form Regarding the Research Process | 12 weeks
  It is a questionnaire formed by the researcher considering the research process and practices and prepared with the opinion of four experts. in form; about the general process of the research, the approach of the interviewer, the approach of the researcher, the training program, the training booklet, the counseling program, the application of guided imagery and its applicability; There are 9 questions that include the feedback of the individuals participating in the research. The form will be applied to the individuals in the experimental group after the post-test data are collected. The feedback of the individuals in the control group will be received after the application of the control group is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Gülnaz Ata, Principal Investigator — Ataturk University
Locations (1):
- Gülnaz Ata, Yakutiye, Erzurum, Turkey (Türkiye)